CLINICAL TRIAL: NCT06538896
Title: Exploratory Single-Arm, Multicenter Phase II Study of Tislelizumab Combined with Nab-Paclitaxel As First Line Treatment for Patients of Triple-negative Breast Cancer(TNBC) with Bone Metastasis
Brief Title: Tislelizumab Combined with Nab-Paclitaxel for First-Line Treatment of Advanced Triple-Negative Breast Cancer with Bone Metastasis，an Exploratory, Single-Arm, Multicenter Phase II Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Hu Hai, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-136
Record Dates: First submitted 2024-07-11; First posted 2024-08-06 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Triple-negative Breast Cancer; Bone Metastases
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — tislelizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab + Nab-Paclitaxel (Experimental): Tislelizumab, 200mg,intravenous, every 3 weeks; nab-paclitaxel, 125mg/m2 on day 1 and day 8, followed by once every three weeks; RANKL inhibitor chosen by investigator is administered at a dose of 120 mg every 4 weeks, with dosing on Days 1, 8, and 15 during the first cycle.
  Interventions: Drug: Tislelizumab + Nab-Paclitaxel; Other: Rankl inhibitor

INTERVENTIONS:
Drug: Tislelizumab + Nab-Paclitaxel — Tislelizumab, 200mg, intravenous, every 3 weeks
Other: Rankl inhibitor — RANKL inhibitor determined by investigator is administered at a dose of 120 mg every 4 weeks, with dosing on Days 1, 8, and 15 during the first cycle.

SUMMARY:
The goal of this clinical trial is to learn if Tislelizumab Combined with Nab-Paclitaxel works to treat patients of TNBC with bone metastasis as first line treatment. It will also learn about the safety of the combination. The main questions it aims to answer are:

How effective is the combination therapy of tislelizumab and nab-paclitaxel in treating advanced first-line triple-negative breast cancer with bone metastasis? And is it safe?

Participants will:

* Receive the treatment as follows: Tislelizumab, 200mg, intravenous, every 3 weeks; nab-paclitaxel, 125mg/m2 on day 1 and day 8, followed by once every three weeks; RANKL inhibitor chosen by investigator is administered at a dose of 120 mg every 4 weeks, with dosing on Days 1, 8, and 15 during the first cycle.
* Visit the clinic once every 3 weeks for checkups and tests
* Keep a diary of their symptoms and the number of times they use a rescue inhaler

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥18 years and <70 years;
2. Metastatic triple-negative breast cancer (TNBC) confirmed by histological examination, i.e., negative for human epidermal growth factor receptor 2 (HER2), estrogen receptor (ER), and progesterone receptor (PR);
3. Eastern Cooperative Oncology Group (ECOG) performance status score: 0-1;
4. Expected survival time ≥3 months;
5. ≥1 bone metastasis confirmed by histology or imaging. There must be at least one measurable lesion defined according to RECIST 1.1 criteria. For lesions that have undergone previous radiotherapy, they can only be considered measurable if there is definite disease progression after radiotherapy;
6. Patients with initially diagnosed stage IV (staging based on AJCC 8th edition) or recurrent/metastatic TNBC who are not suitable for surgical treatment, and have not received prior systemic therapy for advanced disease. Prior neoadjuvant and/or adjuvant therapy with taxanes and other antitumor treatments is allowed, but it must meet the criteria of no progression after neoadjuvant therapy, and the time interval between the end of taxane (neo)adjuvant therapy and recurrence/metastasis must be ≥12 months, and the time interval between the end of capecitabine (neo)adjuvant therapy and recurrence/metastasis must be ≥6 months. If immunotherapy was conducted during neoadjuvant phase, the time interval between the last immunotherapy and the screening enrollment for this study must be ≥24 months;
7. Prior local radiotherapy for metastatic sites is allowed, with no limit on the time of completion of radiotherapy, but the patient must have recovered from the effects of radiotherapy before enrolled;
8. Function of vital organs meets the protocol requirements within 1 week before the first administration of the study drug;
9. Patients voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Currently participating in other clinical studies;
2. Untreated central nervous system disease (patients with asymptomatic central nervous system metastases are allowed);
3. Carcinomatous meningitis;
4. Uncontrolled pleural effusion, ascites, or pericardial effusion (patients with indwelling drainage tubes are allowed to enroll);
5. Existing neuropathy ≥ Grade 2 according to the Common Terminology Criteria for Adverse Events (CTCAE v5.0);
6. Uncontrolled tumor-related pain; patients requiring analgesia are allowed to enroll if they have a stable and effective analgesia regimen at the time of enrollment;
7. Patients expected to use any other systemic or local anti-tumor therapy during the study treatment; local radiotherapy for symptomatic isolated lesions or isolated brain metastases is allowed after evaluation and approval by the investigator; local radiotherapy is not allowed for all target lesions during the study treatment;
8. Diagnosis of other malignancies within 5 years. Exceptions include: radically treated early-stage malignancies (carcinoma in situ or stage I tumors), such as adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer;
9. Currently pregnant/lactating women;
10. Evidence of significant comorbidities that may affect the patients' compliance with the study protocol or interpretation of the study results;
11. Severe cardiovascular disease;
12. Known allergy to any drug used in the study;
13. Patients with any active autoimmune disease requiring systemic treatment (i.e., use of disease-modulating drugs, corticosteroids, or immunosuppressive drugs) within the past 2 years (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; patients with autoimmune-related hypothyroidism receiving stable doses of thyroxine replacement therapy and patients with controllable type 1 diabetes receiving stable doses of insulin are allowed; patients with vitiligo or childhood asthma that has completely resolved and requires no intervention in adulthood are allowed; patients with asthma requiring medical intervention with bronchodilators are not allowed). Replacement therapy (such as thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered systemic treatment;
14. Active hepatitis B patients (including chronic or acute, defined as HBsAg positive at baseline). Previously active HBV infection or cured hepatitis B patients are allowed to enroll if they meet the following conditions: viral hepatitis patients with HBcAb positive and HBsAg negative, with HBV DNA copy number less than the upper limit of normal value of the testing laboratory at the research center before enrollment;
15. Active hepatitis C patients. HCV antibody-positive patients are allowed to enroll only if HCV RNA test results are negative;
16. Other liver diseases with known clinically significance, including alcoholic hepatitis or other hepatitis, cirrhosis, hereditary liver diseases;
17. Known history of HIV positivity or acquired immune deficiency syndrome (AIDS);
18. Prior receipt of allogeneic stem cell or solid organ transplantation;
19. Patients with active tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year before screening;
20. Received systemic immunosuppressive drug treatment within 4 weeks before the first administration of the study drug (including but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF]-α drugs). Patients receiving short-term, low-dose systemic immunosuppressive drug treatment or a single bolus of systemic immunosuppressive drugs (e.g., glucocorticoids for 48 hours to treat contrast allergy) may be enrolled in the study after approval by the medical monitor. Patients receiving mineralocorticoids (such as fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study;
21. Any other severe medical condition or abnormal clinical laboratory results that may hinder the patient's safe participation and completion of the study，based on the investigator's judgment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Up to approximately 33 months
  Objective Response Rate (ORR) - percentage of patients with at least one investigator-assessed visit response of complete or partial response (as assessed by the investigator, using RECIST 1.1)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | The time from date of randomization to the date of progression or death due to any cause, whichever occurs earlier, up to approximately 33 months
  Progression-Free Survival by investigator assessment (in accordance with RECIST 1.1)
Overall Survival (OS) | The time from date of enrollment to the date of death due to any cause up to approximately 33 months
  Overall Survival (OS)
Skeletal Related Events(SRE) | Time from the date of first medication to the first occurrence of pathological fractures, bone surgery, bone radiotherapy, or spinal cord compression caused by tumor bone metastasis, up to 33 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided